CLINICAL TRIAL: NCT01033812
Title: A Pilot Study to Identify and Describe the Male Sexual Partners of Adolescent and Young Adult Women Enrolled in ATN 067
Brief Title: ID & Testing in Male Partners
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 084
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2016-03

CONDITIONS: HIV
Keywords: Networks; Index recruiter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Index Recruiter: Young African American or Latina women who served as index recruiters in ATN 067 and members of their female friendship network members who tested HIV positive based on HIV screening and a confirmatory test result that was conducted in ATN 067.
- Male Sexual Partners: Any male partner who engaged in at least one episode of oral, vaginal or anal sex during the course of their lifetime with an 084 index recruiter.

SUMMARY:
This pilot study is a sub-study of ATN 067. ATN 067 utilizes a cross-sectional research design to recruit Latina and African American young women to undergo HIV screening. The primary goal of this proposed pilot study, ATN 084, is to explore the feasibility and acceptability of index female recruiters identifying and recruiting their past and present male sexual partners to undergo HIV screening and complete a one-time ACASI interview. In addition, the study will also include female friendship network members who were enrolled in ATN 067 and were diagnosed with HIV. These young women will also be asked to recruit their past and present male sex partners to undergo HIV screening.

ELIGIBILITY:
Inclusion Criteria for 084 Index Recruiters:

* 1) Completed participation or is currently enrolled as an index recruiter in ATN 067 or 2) Is a female friendship network member enrolled in ATN 067 who is diagnosed as being HIV infected during her participation in the ATN 067 study;
* Aged 18 years or older at the time of consent;
* Willing to recruit at least one, but no more than six past or current male sexual partners who are willing to discuss and consider HIV screening. A male sexual partner includes individuals with whom the index recruiter has engaged in at least one episode of oral, vaginal or anal sex in the course of their lifetime;
* Able to understand written and spoken English; and
* Willing to provide written informed consent/assent.

Exclusion Criteria for 084 Index Recruiters:

* Self-report of pregnancy at enrollment (pregnancy testing is not required);
* Untreated psychiatric disorder associated with a thought disorder, hallucinations or acute substance use withdrawal. Stabilized patients receiving appropriate psychiatric care will not be excluded if informed consent can be reasonably assumed;
* Visibly distraught and/or visibly emotionally unstable (e.g., depressive mood or exhibiting manic, suicidal, or violent behavior);
* Active drug or alcohol use or dependence that, in the opinion of the site personnel, would interfere with ability to give true informed consent and adhere to the study requirements or;
* Acute illness that, in the opinion of the treating clinician, would interfere with the participant's ability to adhere to the protocol requirements and/or interfere with the protocol objectives.

Inclusion Criteria for Male Sexual Partners:

* Is born male;
* Aged 18 years or older at the time of consent;
* Identified as a male sexual partner of an index recruiter enrolled in ATN 067 (having had vaginal and/or anal sexual intercourse in the past);
* Willing to complete a sociodemographic and behavioral risk assessment survey;
* Willing to discuss and consider HIV screening;
* Able to understand written and spoken English; and
* Willing to provide written informed consent/assent.

Exclusion Criteria for Male Sexual Partners:

* Untreated psychiatric disorder associated with a thought disorder, hallucinations, and/or acute substance use withdrawal. Stabilized patients receiving appropriate psychiatric care will not be excluded if informed consent can be reasonably assumed;
* Visibly distraught and/or visibly emotionally unstable (e.g., depressive mood or exhibiting manic, suicidal, or violent behavior);
* Active drug or alcohol use or dependence that, in the opinion of the site personnel, would interfere with ability to give true informed consent and adhere to the study requirements or;
* Acute illness that, in the opinion of the treating clinician, would interfere with the participant's ability to adhere to the protocol requirements and/or interfere with the protocol objectives.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will include index recruiters and their male sexual partners. The index recruiters will be comprised of young women who served as index recruiters in ATN 067 and members of their female friendship network members who tested HIV positive based on HIV screening and a confirmatory test result that was conducted in ATN 067. All study participants will be 18 years of age or older.
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To examine the feasibility of identifying/recruiting the male sex partners of African American and Latina sexually experienced females aged 18 or older who were either index recruiters in ATN 067 or their HIV-infected female friendship network members. | 2 months
To conduct HIV screening among the male sexual partners of the ATN 084 female index recruiters and examine factors that facilitate and hinder these individuals in undergoing HIV screening. | 2 months

SECONDARY OUTCOMES:
To compare sociodemographic characteristics, risk behaviors, psychosocial variables and self-reported sex partners of the male sexual partners of the ATN 084 female index recruiters. | 2 months
To describe sexual mixing patterns (assortative/dissortative), bridging and concurrency among the ATN 084 index recruiters and their male sexual partners by age race/ethnicity and HIV status. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hightow-Weidman, M.D., MPH, Study Chair — Adolescent Trials Network; Cherrie Boyer, Ph.D., Study Chair — Adolescent Trials Network
Locations (3):
- United States (3):
  - University of Miami School of Medicine, Miami, Florida
  - Ruth M Rothstein CORE Center/ John H Stroger Jr Hospital, Chicago, Illinois
  - Montefiore Medical Center, The Bronx, New York

REFERENCES:
- See also: ATN Website — http://www.atnonline.org